CLINICAL TRIAL: NCT00791284
Title: Pharmacokinetics of Paliperidone in Subjects With Moderate Hepatic Impairment as Compared to Subjects With Normal Hepatic Function.
Brief Title: A Study of the Pharmacokinetics of Paliperidone in Volunteers With Normal or Impaired Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004204
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia; Hepatic Impairment
Keywords: Schizophrenia; Mood disorders; Antipsychotic drugs; intermediate release (IR) Paliperidone
MeSH Terms: conditions — Schizophrenia; Mood Disorders | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: Intermediate release (IR) Paliperidone

SUMMARY:
The purpose of this study is 1) to investigate the single-dose pharmacokinetics of immediate release (IR) paliperidone, after oral administration, in patients having moderate hepatic impairment compared to patients having normal hepatic function, 2) to document the plasma protein binding and disposition of the enantiomers of paliperidone, and 3) to evaluate the tolerability and safety profile of IR paliperidone in both patient populations.

DETAILED DESCRIPTION:
This is a single-dose, parallel-group, open-label, single-center, Phase 1 study of immediate release (IR) paliperidone in patients having either normal or moderately-impaired hepatic function. The groups, which will consist of 10 patients each, will be demographically matched with respect to age, weight, sex, and ethnicity. The study will consist of a screening period of up to 3 weeks and an open-label, single-dose treatment period (Days 1 through 5). On Day 1, a single dose of 1 mg Intermediate Release (IR) paliperidone oral solution will be administered after a fast of at least 10 hours; patients will continue to fast for 4 hours following study drug administration. The 96-hour follow-up will consist of serial sample collections of blood and urine for pharmacokinetic analysis and safety and tolerability assessments. Patients will remain confined to the study site through the 72-hour pharmacokinetics sampling and will consume standard institutional meals while in the study site. Patients will be released after the 72-hour sampling, then will return to the study site on Day 5 before the 96-hour pharmacokinetics sampling; end-of-study procedures will be performed immediately thereafter. Currently, pharmacokinetic data are available after oral IR and Extended Release (ER) formulations of paliperidone were administered to healthy patients and to patients with schizophrenia who had normal hepatic function. No pharmacokinetic information on paliperidone in patients with hepatic impairment has been obtained. The target population for paliperidone comprises schizophrenic patients. Because some patients in the target population might be hepatically impaired, pharmacokinetic information in this population is helpful. This single-dose pharmacokinetic study will collect information in patients with normal hepatic function and in patients with moderate hepatic impairment to provide clinical dosing information/recommendations for patients with hepatic impairment. Safety and tolerability will be monitored. A single dose of 1 mg intermediate release (IR) paliperidone oral solution

ELIGIBILITY:
Inclusion Criteria:

* Patients with normal hepatic function:Normotensive at screening, with supine (5 minutes) blood pressure between the range of 95 to 160 mmHg systolic, inclusive, and 55 to 95 mmHg diastolic, inclusive, demographically comparable to the hepatic impairment group with respect to age, weight, sex, and ethnicity and healthy on the basis of a prestudy physical examination, medical history, ECG, and laboratory results of blood biochemistry, hematology, and urinalysis performed within 3 weeks before study drug administration. If the results of the biochemistry or hematology tests or the urinalysis are not within the laboratory's reference ranges, the patient can be included only if the investigator judges that the deviations are not clinically significant
* Patients with moderate hepatic impairment: Blood pressure controlled and stable on antihypertensive agents, stable hepatic disease with laboratory and clinical findings that support the diagnosis of hepatic impairment, otherwise healthy on the basis of a prestudy physical examination, medical history, ECG, and laboratory results of blood biochemistry, hematology, and urinalysis performed within 3 weeks before study drug administration. Patients with controlled hypertension and those problems directly associated with the primary diagnosis of hepatic impairment may be included. Patients with stable, mild, chronic concurrent diseases, such as degenerative joint disease, Type II diabetes, or thyroid conditions requiring thyroid replacement therapy or surgery, may be included. If the results of the biochemistry or hematology tests or the urinalysis are not within the laboratory's references ranges, the patient can be included only if the investigator judges that the deviations are not clinically significant. Laboratory results related to the patient's underlying condition may be outside of the normal ranges. (Serum bilirubin, albumin, and prothrombin time will be assessed individually)
* Total score of Child-Pugh's classification will be between 7 and 9, inclusive
* Concomitant medications to treat underlying disease states or medical conditions related to hepatic insufficiency are allowed. Patients have to be on a stable dose of medication and/or treatment regimen 2 months before the study, as well as during the study.

Exclusion Criteria:

* Patients with normal hepatic function:Has any significant history or presence of hepatic disease or has positive serology result for hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus (as determined by a multi-antigen enzyme immunoassay)
* At screening, sustained drops in systolic (>20 mmHg) or diastolic (>10 mmHg) blood pressure after standing for at least 2 minutes which are not associated with an increase in pulse rate of >15 beats per minute
* Is taking, or has taken, any prescribed or over-the-counter drug (including vitamins and herbal supplements) within 2 weeks before study drug administration (with the exception of paracetamol, hormonal contraceptives, and hormone replacement therapy)
* Patients with moderate hepatic impairment: Has any clinically significant laboratory abnormality except those parameters influenced by hepatic impairment, has a score of 3 or 4 for hepatic encephalopathy as determined by the result of the Number Connection Test, has severe ascites and/or pleural effusion, has serology result positive for HBsAg, has acute exacerbation of liver disease, as indicated by worsening clinical signs of hepatic impairment, or by an increase of more than 50% in total bilirubin or prothrombin time in the preceding 3 months (as far as information is available).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-08; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
To investigate the single-dose pharmacokinetics of IR paliperidone after oral administration to patients with moderate hepatic impairment as compared to patients with normal hepatic function

SECONDARY OUTCOMES:
To document the plasma protein binding and disposition of the enantiomers of paliperidone and to evaluate the tolerability and safety profile of IR paliperidone in both patient populations

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the pharmacokinetics of paliperidone in volunteers with normal or impaired liver function — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=566&filename=CR004204_CSR.pdf